CLINICAL TRIAL: NCT04747847
Title: Pilot Study of Atorvastatin and Anakinra in Children With Coronary Artery Abnormalities Secondary to Kawasaki Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Adriana H. Tremoulet, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD Combo; R01HL140898 (NIH)
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Atorvastatin; Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atorvastatin and anakinra (Experimental): Anakinra up to 8 mg/kg/day and atorvastatin at 0.75 mg/kg/day
  Interventions: Drug: Atorvastatin and anakinra

INTERVENTIONS:
Drug: Atorvastatin and anakinra — Anakinra up to 8 mg/kg/day and atorvastatin at 0.75 mg/kg/day in children with acute KD at least 1 year old with CAA

SUMMARY:
Kawasaki disease (KD) is the leading cause of acquired heart disease in children in the developed world. Despite available treatment, 25% of children in San Diego County appropriately treated for KD develop coronary artery abnormalities that could lead to complications later in life, including heart attack. Although we can identify children with KD that have these coronary artery abnormalities, there is no approved additional treatment to decrease coronary artery inflammation and arrest or prevent damage to the coronary arteries. Statins, a class of drugs that is known for lowering cholesterol, have also been shown to decrease inflammation in general as well as at the level of the vessel wall. Anakinra, a therapy that blocks the high levels of interleukin 1 (IL1) that leads to inflammation during acute KD, has been shown in the KD mouse model to prevent the development of coronary artery damage. Both of these therapies have been demonstrated to be safe and well-tolerated in KD patients. Therefore, we propose to study the effects of combination therapy with atorvastatin and anakinra in children with acute KD and early coronary artery abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Acute Kawasaki disease with a Z score of 3 or larger of the LAD or RCA

Exclusion Criteria:

* Taking a CYP3A4 metabolized drug (such as cyclosporine)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 6 weeks
  The number of participants with adverse events related to study drugs will be assessed and reported

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Tremoulet, MD, Principal Investigator — Professor
Locations (1):
- University of California San Diego, San Diego, California, United States